CLINICAL TRIAL: NCT03955029
Title: Effects of Progressive Interval Training on V02 Max in Chronic Heart Failure Patients
Brief Title: Interval Training in Heart Failure
Acronym: PROVO2MAX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RECHMPL18_0229
Record Dates: First submitted 2019-04-05; First posted 2019-05-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Interval training (Experimental): It is a split-type workout that alternates periods of intensity between 60% -95% of the maximum effort (depending on the modality) and periods of passive or active rest between 20-30% of the maximum effort. The experimental group will follow conventional Interval Training
  Interventions: Other: Conventional Interval training
- Progressive Interval training (Experimental): It is a split-type workout that alternates periods of intensity between 60% -95% of the maximum effort (depending on the modality) and periods of passive or active rest between 20-30% of the maximum effort. The experimental group will follow progressive Interval Training
  Interventions: Other: Progressive Interval training

INTERVENTIONS:
Other: Progressive Interval training — heating up 7 minutes at 15 watt, then alternating 30% of the maximum power reached by the patient at Vo2 max for 3 minutes and first peak at 40% of max power, second at 45%, third at 50%, fourth at 55 % and fifth to 60%, then return to calm 3 minutes at 15 watt. Total duration of the endurance session: 30 minutes. The powers of the peak will be modeled according to the Borg (if <6, increase by 5 watt the value of each peak at the next session).
  Arms: Progressive Interval training
Other: Conventional Interval training — warm up 7 minutes at 15 watt, then alternating between plateau at 30% of the max power reached by the patient at VO2 max for 3 minutes and peak at 60% for 1 minute, return to calm 3 minutes at 15 watts. Total duration of the endurance session: 30 minutes. The power of the peak will be modeled according to the Borg (if <6, increase by 5 watt the value of each peak at the next session)
  Arms: Conventional Interval training

SUMMARY:
Heart failure (HF) is currently considered a common pathology, with 15 million adults in Europe and 26 million worldwide. The American Heart Association (AHA) estimates that their number will increase by 25% by 2030. In France, HF affects more than one million people. Because of the repeated hospitalizations of this disease, it is considered a costly pathology and with a high mortality rate (23.000 deaths per year in France). Moreover, HF is a severe pathology that affects the quality of life of patients and their families. Treatment and medical follow-up are required.

A cardiac rehabilitation program is also a primary indication according to the latest recommendations and repositories in Cardiology. Various studies show that "Interval Training" exercise program improves VO2 peak compared to a "continuous" program, which constitutes a major prognostic factor in the population of heart failure. However, it is sometimes a difficult program to offer to more deconditioned patients as it requires reaching powers around 80% - 95% of its maximum exertion capacity. So, a variant of the interval training is offered, called Progressive Interval Training (PIT), based on the same model as the conventional interval training (CIT), but with an increasing power and breathing threshold, so that the patient can adapt gradually.

The hypothesis is that PIT could improve VO2 peak better than CIT in cardiac rehabilitation program. Therefore, study the benefits of PIT training to improve the conditioning and quality of life of patients with chronic heart failure will be studied.

DETAILED DESCRIPTION:
Chronic Heart Failure (CHF) is due to structural or functional cardiac anomalies which causes a lack of oxygen perfusion to various organs provoking symptoms as dyspnea, fatigue, palpitation at rest or during efforts. International prevalence is 1-2% in adult population, wich represents 15 million people in Europe and 26 millions in the world. In France, CHF represents the first cause of hospitalization. The rate of intra-hospital mortality is 8.2 % and the mortality in 1 year is 26 % according to the study OFICA in 2013. Its treatment is first medication.

Cardiac rehabilitation programs are also proposed. According to the latest recommendations of the European Society of Cardiology in 2016, patient education on diet, medical treatment observance and facilitation of psychosocial assistance with access to a multidisciplinary team, will reduce the rate of hospitalization and mortality (level of evidence IA). Similarly, the regular practice of an aerobic-type activity will increase the patient's functional capacity and improve the symptoms related to the disease. In the same way, the risk of re-hospitalization will be reduced (level of evidence IA). Cardiac rehabilitation of CHF patients includes a so-called "segmentary analytics" rehabilitation based on strength exercises and aerobic-type endurance work. This classical program is called "continuous" training in which the patient must exert on a cycloergometer or walking on a treadmill between 60% and 70% of his maximum exertion capacity, evaluated with initial VO2 max exercise test, before cardiac rehabilation. More recently, a new form of rehabilation mode appeared: "Interval Training" (IT) inspired by high level athletes training. It is a training model that alternates periods of intensity between 60%-95% of maximum effort (depending on the modality) and periods of passive or active rest between 20-30% of maximum effort. IT is more suitable for endurance work in CHF patients than continuous training. Indeed, this type of exercise has a muscular impact, in terms of strength, superior to that brought by continuous training without significantly increasing cardiac work or hemodynamic and metabolic parameters. Some studies show the effectiveness of both types of programms (continuous or IT) on improving the 6 minute walk test distance (6MWD) and displacing the first ventilatory threshold (VT1) for higher intensities. However, the interval training has a better effect than continuous program: 19.4% versus 8.3% for 6MWD improvement and 95% versus 75% for heart peak rate gain.

Nevertheless, it have been observed in daily practice that classical conventional IT (CIT) program could be difficult to perform in most of CHF patients, due to the severity of their pathology, poor physical condition and especially muscle deconditioning. Indeed, this deconditioning is linked to the sedentary behaviour of this type of patient because of the specific symptoms of his cardiac pathology, which will result in severe intolerance to effort. In Cardiac rehabilitation department of Montpellier University Hospital, a new type of IT program for severe CHF patients have been tested, with progressive intervals of maximum effort and active rest periods, called the Progressive Interval Training (PIT) program. After 6 months of applying this training model to our patients, it seems to be effective in endurance gain in final exercise test and without side-effects in terms of safety. The objective is to compare the 2 types of IT workouts (CIT and PIT) in 2 different randomized groups, on the improvement of VO2 peak in patients with severe CHF. Secondary ojectives are the imporvemnt on 6MWD, life quality and ventilatory threshold at the end of rehabilitation (VT1).

A typical session for a patient takes place in two parts: the first one with analytical segmentary rehabilitation exercises identical in terms of the muscular group worked and the number of series and repetitions and adapted (charge in kg) to each patient, and a second one of endurance aerobic work with conventional interval training (CIT) program or progressive interval training (PIT) program according to the randomized groups.

* CIT intervention consists in: warming 7 minutes at 15 watts, then alternating exercices phases at 30% of maximum power (reached by patient at initial VO2 maximal exercise test realized before cardiac rehabilation) during 3 minutes and peak at 60% of maximum watts during 1 minute, then return to calm 3 minutes at 15 watts. Total duration of the endurance session is 30 minutes. The power in watts of the peak work will be shaped according to the Borg (if 6, increase of 5 watt the value of each peak at the next session).
* PIT intervention consists in: warming 7 minutes at 15 watts, then alternating exercices phases at 30% watts of maximum power (reached by patient at initial VO2 maximal exercise test realized before cardiac rehabilation) during 3 minutes, a first peak work at 40% of maximum power, a second at 45%, a third at 50%, a fourth at 55% and a fifth at 60%, then return to calm 3 minutes at 15 watts. Total duration of this endurance session is also 30 minutes. The peak powers will be shaped according to the Borg (if 6, increase of 5 watt the value of each peak to the next session).

Each patient conducts a total of 20 sessions at a rate of 2 sessions per week. It is a monocentric, controlled, randomized, prospective study with two parallel groups (open except for the evaluation which will be blind). The sample size is estimated at 50 subjects. Inclusion criteria are patients with CHF (left ventricular ejection fraction <40%), men or women over 60 years of age, admitted on a cardiac rehabilation medical, with a functional capacity of less than 5 Mets, all of whom have their free and informed consent for the study.

The benefits to the patient are those related to Cardiovascular Rehabilitation that increase its functional capacity while improving its quality of life.

If the effectiveness of PIT program on improving aerobic capacity (VO2 max), functional abilities (VT1, TDM6 ') and/or quality of life is demonstrated, this program could be recommended for cardiac rehabilitation in patients with severe CHF. A larger number of patients could benefit from this program which takes into account the muscular deconditioning related to their pathology.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic systolic heart failure (LVEF <40%)
* men or women
* 40 years patients or older
* Patients admitted on cardiac rehabilitative medical prescription
* Patients with a functional capacity of 6 Mets or less
* Patients having given their free and informed consent to the study.

Exclusion Criteria:

* Contraindication to rehabilitation,
* Refusal of the patient to participation in the study
* impaired comprehension
* inability to perform the cyclometer
* participation in another therapeutic protocol simultaneously

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-01-10 (Actual); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-01-10 (Estimated)

PRIMARY OUTCOMES:
VO² peak in patients with cardiac heart failure | Baseline
  Evaluate the effectiveness of endurance rehabilitation program with climbing of ladders (PIT) versus an endurance rehabilitation program with conventional interval training on improving VO² peak in patients with CHF
VO² peak in patients with cardiac heart failure | 12 weeks
  Evaluate the effectiveness of endurance rehabilitation program with climbing of ladders (PIT) versus an endurance rehabilitation program with conventional interval training on improving VO² peak in patients with CHF

SECONDARY OUTCOMES:
Questionnary Short Form Health Survey | Baseline
  Questionnary Short Form Health Survey (SF-36)
Questionnary Short Form Health Survey | 12 weeks
  Questionnary Short Form Health Survey (SF-36)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided